CLINICAL TRIAL: NCT02699385
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group, Prospective Study to Evaluate the Safety and Efficacy of Domperidone in 6-month-old to 12-year-old Pediatric Subjects With Nausea and Vomiting Due to Acute Gastroenteritis
Brief Title: A Study to Evaluate the Safety and Efficacy of Domperidone in Pediatric Participants With Nausea and Vomiting Due to Acute Gastroenteritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study prematurely terminated upon recommendation of IDMC due to lack of efficacy.
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107501; R033812GTS3001 (Other: Janssen-Cilag International NV); 2015-002923-24 (EudraCT Number)
Record Dates: First submitted 2016-02-15; First posted 2016-03-04 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Gastroenteritis
Keywords: Gastroenteritis; Domperidone; Pediatric participants
MeSH Terms: conditions — Gastroenteritis | interventions — Fluid Therapy; Domperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Rehydration Therapy (ORT) + Domperidone (Experimental): Each participants will initiate ORT in the physician's office and domperidone 0.25 milligram per kilogram (mg/kg) of body weight of oral suspension thrice daily for up to 7 days.
  Interventions: Other: Oral Rehydration Therapy; Drug: Domperidone
- Oral Rehydration Therapy + Placebo (Experimental): Each participants will initiate ORT in the physician's office and placebo oral suspension thrice daily for up to 7 days.
  Interventions: Other: Oral Rehydration Therapy; Drug: Placebo

INTERVENTIONS:
Other: Oral Rehydration Therapy — Each participants will initiate ORT in the physician's office on Day 1.
Drug: Domperidone — Each participants will receive Domperidone 0.25 milligram per killogram (mg/kg) of body weight of oral suspension thrice daily for up to 7 days.
  Arms: Oral Rehydration Therapy (ORT) + Domperidone
Drug: Placebo — Each participants will receive placebo oral suspension thrice daily for up to 7 days.
  Arms: Oral Rehydration Therapy + Placebo

SUMMARY:
The purpose of this study is to demonstrate that domperidone suspension plus oral rehydration therapy (ORT) is more effective than placebo plus ORT at reducing the symptoms of vomiting associated with acute gastroenteritis (AG) within the first 48 hours of treatment administration in pediatric participants with AG and mild-to-moderate dehydration.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), double-blind (neither the researchers nor the participants know what treatment the participant is receiving), parallel-group, placebo-controlled, multicenter (when more than one hospital or medical school team work on a medical research study) study. The study consists of 3 Phases: Screening Phase (-2 to 0 hours prior to baseline on Day 1), Double-blind treatment Phase (up to 7 Days) and follow-up Phase (7 Days). The duration of participation in the study for each participant is at most 15 Days. Efficacy and safety of domperidone will be evaluated. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* The participant presents with at least 3 episodes of non-bilious, non-bloody vomiting within the 24 hours prior to visiting the physician's office. The participant has at least 2 signs and symptoms other than vomiting consistent with acute gastroenteritis (AG) (example, fever, nausea, diarrhea, abdominal pain, bloating, or discomfort) within 3 hours prior to visiting the physician's office
* The participant has mild-to-moderate dehydration
* The participant had at least 1 episode of non-bloody diarrhea within the 24 hours prior to the visiting the physician's office

Exclusion Criteria:

* The participant has severe dehydration or severe malnutrition
* The participant who has vomiting and clinical symptoms for longer than 72 hours prior to the baseline physician's office visit
* The participant needs intravenous (IV) fluid replacement
* The participant has chronic severe diarrhea, a previous history of Helicobacter pylori infection or received treatment for H. pylori-induced gastritis, active peptic ulcer, celiac disease, Crohn's disease, ulcerative colitis, eosinophilic esophagitis, malabsorption, short bowel syndrome, post-viral gastroparesis, cyclic vomiting syndrome, or previous gastrointestinal surgery
* The participant has upper respiratory symptoms such as cough, congestion, otitis media or pharyngitis

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With No Vomiting Episode Within the First 48 Hours of the First Treatment Administration | 48 Hours
  The vomiting episodes will be recorded for each participants in the eDiary.

SECONDARY OUTCOMES:
Percentage of Participants 4 Years of Age or Older Who Have No Episode of Nausea Within the First 48 Hours of the First Treatment Administration | 48 Hours
  The nausea episodes will be recorded in the eDiary.
Number of Vomiting Episodes for Participants Within the 0 to 24 Hour, Greater Than (>) 24 to 48 Hour, and >48 Hour to 7 Day Periods After the First Treatment Administration | Up to Day 7
  The vomiting episodes will be recorded for each participants in the eDiary.
Number of Episodes of Nausea for Participants 4 Years of Age or Older Within the 0 to 24 Hour, >24 to 48 Hour, and >48 Hour to 7 Day Periods After the First Treatment Administration | Up to Day 7
  The nausea episodes will be recorded in the eDiary.
Percentage of Participants who Have No Episode of Vomiting Within the 0 to 24 Hour, >24 to 48 Hour, and >48 Hour to 7 Day Periods After the First Treatment Administration | Up to Day 7
  The vomiting episodes will be recorded for each participants in the eDiary.
Percentage of Participants 4 Years of Age or Older Who Have No Episode of Nausea Within the 0 to 24 Hour, >24 to 48 Hour, and >48 Hour to 7 Day Periods After the First Treatment Administration | Up to Day 7
  The nausea episodes will be recorded in the eDiary.
Percentage of Participants Who Have No Episode of Vomiting Within the 7 Day Treatment Period After the First Treatment Administration | Day 7
  The vomiting episodes will be recorded for each participants in the eDiary.
Percentage of Participants 4 Years of Age or Older Who Have No Episode of Nausea Within the 7 Day Treatment Period After the First Treatment Administration | Day 7
  The nausea episodes will be recorded in the eDiary.
Percentage of Participants Taking a Rescue Medication Within the 7 Day Treatment Period | Day 7
  If nausea, vomiting, or diarrhea worsens during the study and the investigator initiates rescue medication, the study medication will be discontinued.
Percentage of Participants Stopping Study Medication Early Due to Vomiting-Free for 24 Hours Within the 7 Day Treatment Period | Day 7
  The vomiting episodes will be recorded for each participants in the eDiary.
Time to Last Study Medication Within the 7 Day Treatment Period | Day 7
  Time taken to administer last study medication will be observed.
Percentage of Participants Referred to an Emergency Room/Hospital for Treatment Within the 7 Day Treatment Period | Day 7
  If nausea, vomiting, or diarrhea worsens during the study and admits the participant to the hospital for IV fluids, the study medication will be discontinued.
Time-to-Last Vomiting Within the 7 Day Period After the First Treatment Administration | Day 7
  The vomiting episodes will be recorded for each participants in the eDiary.
Change From Baseline in Hydration Score at Day 2 | Baseline and Day 2
  The severity of dehydration will be assessed using the Dehydration Score Assessment. a) Children under 24 months of age with a score range 7 to 10 points have mild dehydration and children with a score range of 11 to 17 points have moderate dehydration (only children under 24 months of age are evaluated for tears). b) Children 24 months of age or older with a score range of 6 to 9 points have mild dehydration and children with a score range of 10 to 15 points have moderate dehydration. and c) Children under 24 months of age with scores of 18 or more and children 24 months of age or older with scores of 16 or more are considered to be severely dehydrated and are excluded from the study.
Change From Baseline in Weight at Day 2 | Baseline and Day 2
  Weight will be measured to the nearest 100 grams in underwear (no diaper/nappy/training pants).
Percentage of Participants With Diarrhea Within 0 to 24 Hour, >24 to 48 Hour, >48 Hour to 7 Day, and 0 Hour to 7 Day Periods After the First Successful Treatment Administration | Up to Day 7
  The diarrhea episodes will be recorded for each participant in the eDiary.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (29):
- Austria (3):
  - Gröbming
  - Salzburg
  - Vienna
- Belgium (4):
  - Brussels
  - Herbeumont
  - Massemen
  - Moorsel
- Russia (2):
  - Novosibirsk
  - Saint Petersburg
- South Africa (7):
  - Cape Town
  - Durban
  - Krugersdorp
  - Middelburg
  - Newtown
  - Pietermaritzburg
  - Pretoria
- Spain (4):
  - Burriana
  - Gandia
  - Valencia
  - Vic
- United Kingdom (9):
  - Barnsley
  - Ipswich
  - Maidstone
  - Middlesbrough
  - Nottingham
  - Oldham
  - Royal Tunbridge Wells
  - Staffordshire
  - Sutton in Ashfield

REFERENCES:
- [Derived] Leitz G, Hu P, Appiani C, Li Q, Mitha E, Garces-Sanchez M, Gupta R. Safety and Efficacy of Low-dose Domperidone for Treating Nausea and Vomiting Due to Acute Gastroenteritis in Children. J Pediatr Gastroenterol Nutr. 2019 Oct;69(4):425-430. doi: 10.1097/MPG.0000000000002409. PMID 31181017
- See also: A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group, Prospective Study to Evaluate the Safety and Efficacy of Domperidone in 6-month-old to 12-year-old Pediatric Subjects With Nausea and Vomiting Due to Acute Gastroenteritis — https://www.clinicaltrialsregister.eu/ctr-search/trial/2015-002923-24/results